CLINICAL TRIAL: NCT00031447
Title: A Placebo-Controlled Phase III Evaluation of Suppressive Therapy With Oral Acyclovir Suspension Following Neonatal Herpes Simplex Virus Infections Limited to the Skin, Eye, and Mouth
Brief Title: Acyclovir Herpes Simplex Virus (HSV) Skin, Eye, and Mouth
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 97-006; CASG 104; N01AI30025C; N01AI30025 (NIH); NCT00001099 (obsolete NCT alias)
Record Dates: First submitted 2002-03-06; First posted 2002-03-07 (Estimated); Results first posted 2010-04-09 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2009-11

CONDITIONS: Herpes Simplex
Keywords: Herpes Simplex, Acyclovir, Infants
MeSH Terms: conditions — Herpes Simplex | interventions — Acyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Acyclovir (Experimental)
  Interventions: Drug: Acyclovir

INTERVENTIONS:
Drug: Acyclovir — Oral suspension 300 mg/m^2/dose, 3 times per day (TID), for 6 months.
  Arms: Acyclovir
Drug: Placebo — Placebo identical to oral acyclovir suspension in appearance and taste.
  Arms: Placebo

SUMMARY:
The purpose of this study is to test whether long-term treatment with oral acyclovir improves the outcome for infants with herpes simplex virus (HSV) disease of the skin, eyes, and mouth (SEM). Study participants will include infants in the United States and Canada who have HSV disease of the skin, eyes, and mouth, with no central nervous system disease present. Initially, all subjects will be treated with acyclovir administered through IV access (through the vein) for 14 days while hospitalized. Participants will then be placed in one of two groups, acyclovir given by mouth or a placebo (substance with no medication present). The participant and the study site will not know to which group the subject is assigned. All children will be followed at 6, 12, 24, 36, 48, and 60 months of age. During the follow up visits, physicals, hearing assessments, eye assessments, and neurological assessments will be completed.

DETAILED DESCRIPTION:
Neonatal herpes simplex virus (HSV) disease complicates approximately one in every 3,000 births in the United States. This study will be a placebo-controlled Phase III evaluation of suppressive therapy with oral Acyclovir suspension following neonatal HSV infections limited to the skin, eyes, and mouth (SEM). This study will evaluate the efficacy of long-term suppressive therapy with oral acyclovir in infants with SEM disease. It will determine if suppressive oral acyclovir therapy improves neurological outcome in infants following SEM disease. Only infants with SEM disease will qualify for this study. After qualifying for the study and obtaining informed consent, the infant will complete 14 days of intravenous (IV) Acyclovir (20 mg/kg/dose given every 8 hours). Patients will be randomized to receive suppressive oral Acyclovir versus placebo only if they continue to meet all study inclusion criteria at the completion of the IV therapy. This study will be double-blinded and placebo controlled. At the time of randomization, the patient will be placed in 1 of 2 groups (oral suppressive Acyclovir versus placebo). If a patient in either group has a cutaneous HSV recurrence, open-label oral Acyclovir (80 mg/kg/day divided into 4 doses per day) will be provided for 5 days. During the time of administration of open-label oral Acyclovir, study drug will be withheld. All children will be followed at 6, 12, 24, 36, 48, and 60 months of age. Physical examination, hearing assessment, and retinal examination will be performed at each follow up visit. Standardized neurologic evaluation will be performed at 12, 24, 36, 48, and 60 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Isolation by viral culture of herpes simplex virus (HSV)-1or HSV-2 from cutaneous lesions, conjunctivae, or oropharynx. Detection of HSV at any of these sites is sufficient, and the presence of skin lesions is not required for study enrollment.
* Normal cerebrospinal fluid (CSF) indices (<22 white blood cells (WBCs)/mm^3 and protein <115 mg/dl for term infants; (<25 WBCs/mm^3 and protein <220 mg/dl for preterm infants both at the time of diagnosis of HSV disease and at the time of study randomization.
* No evidence of HSV central nervous system (CNS) disease by computed tomography (CT) with contrast, magnetic resonance imaging (MRI) with gadolinium, or head ultrasound (HUS) [NOTE: CT with contrast is the preferred imaging study].
* Normal electroencephalogram (EEG), if performed [NOTE: EEG is suggested for the evaluation of infants with HSV disease but is not required for this study].
* No evidence of visceral dissemination of HSV infection (normal liver function tests, normal chest x-ray, etc.).
* Negative CSF HSV polymerase chain reaction (PCR) results from specimens obtained both within 72 hours of initiation of intravenous acyclovir therapy and within 48 hours prior to completion of intravenous acyclovir therapy.
* Less than or equal to 28 days of age at the time of initial presentation with skin, eyes, and mouth (SEM) disease.
* Birth weight greater than or equal to equal to 800 grams.

Exclusion Criteria:

* Infants with either grade 3 or grade 4 intraventricular hemorrhage (IVH) prior to study enrollment.
* Breast feeding infants whose mothers are taking acyclovir, valacyclovir, or famciclovir for >120 hours (>5 days). If at any point following enrollment the mother takes these antiviral drugs for >120 hours (>5 days), she will be asked to refrain from breast feeding while taking the drug.
* Infants known to be born to women who are human immunodeficiency virus (HIV) positive (but HIV testing is not required for study entry). These infants are at known risk for acquiring HIV, which would alter their immune response to other infections, including HSV infection. Additionally, they may be receiving antiretroviral and/or antiviral drugs during the time in which the study of suppressive oral acyclovir is being conducted. As such, they will be excluded if the mother's positive HIV status is known at the time of evaluation for study inclusion. If at any point following enrollment it is learned that an infant is HIV positive, he/she will be continued on the study protocol.
* Infants with either central nervous system (CNS) or disseminated HSV infection. Patients with CNS HSV infection will be considered for enrollment and randomization in the ongoing Collaborative Antiviral Study Group (CASG) evaluation of oral suppressive acyclovir therapy following neonatal HSV infections involving the CNS.
* Infants with creatinine >1.5mg/dl at time of study enrollment.
* Infants receiving acyclovir expectantly do not qualify for this study because they never developed HSV disease. Expectant therapy describes infants who are cultured at approximately 24 hours of life because of a risk of HSV infection (i.e. they are born to women with active genital lesions). Oftentimes, if these cultures are positive, the infant will receive a course of intravenous acyclovir to prevent the development of HSV disease. However, since they never actually had HSV disease, their potential outcome cannot be compared with infants with typical skin, eyes, and mouth (SEM) disease, and so they are not included in this study.

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 1999-08; Primary Completion 2008-02 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (27):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arkansas Children's Hospital, Department of Infectious Diseases, Little Rock, Arkansas
  - Rady Children's Hospital San Diego, San Diego, California
  - Stanford University School of Medicine, Stanford, California
  - University of Florida - College of Medicine - Jacksonville, Jacksonville, Florida
  - The University of Chicago - Comer Children's Hospital - Infectious Diseases, Chicago, Illinois
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane University - Tulane Medical Center - Department of Pediatrics, New Orleans, Louisiana
  - Maine Medical Center - Department of Pediatric Specialty Care - Infectious Disease, Portland, Maine
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Children's Hospital of Michigan - Pediatric Infectious Diseases, Detroit, Michigan
  - University of Mississippi, Jackson, Mississippi
  - Washington University School of Medicine in St. Louis - Center for Clinical Studies, St Louis, Missouri
  - Mount Sinai Hospital, New York, New York
  - UNY Upstate Medical University Hospital - Pediatrics, Syracuse, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - MetroHealth Medical Center - Pediatric Infectious Disease, Cleveland, Ohio
  - Nationwide Children's Hospital - Infectious Diseases, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Cook Children's Infectious Disease Services, Fort Worth, Texas
  - University of Texas Health Science Center San Antonio - Pediatrics - Immunology & Infectious Disease, San Antonio, Texas
  - Seattle Children's Hospital - Infectious Diseases, Seattle, Washington
- University of Alberta - Aberhart Centre - Pediatrics, Edmonton, Alberta, Canada

REFERENCES:
- [Result] Kimberlin DW, Whitley RJ, Wan W, Powell DA, Storch G, Ahmed A, Palmer A, Sanchez PJ, Jacobs RF, Bradley JS, Robinson JL, Shelton M, Dennehy PH, Leach C, Rathore M, Abughali N, Wright P, Frenkel LM, Brady RC, Van Dyke R, Weiner LB, Guzman-Cottrill J, McCarthy CA, Griffin J, Jester P, Parker M, Lakeman FD, Kuo H, Lee CH, Cloud GA; National Institute of Allergy and Infectious Diseases Collaborative Antiviral Study Group. Oral acyclovir suppression and neurodevelopment after neonatal herpes. N Engl J Med. 2011 Oct 6;365(14):1284-92. doi: 10.1056/NEJMoa1003509. PMID 21991950

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Neonates diagnosed with HSV-1 or HSV-2 at least than or equal to 28 days of age as evidenced by infections limited to the skin, eye and mouth with normal CNS and treated with intravenous acyclovir therapy.
Pre-assignment Details: Participants enrolled while on 2 weeks of IV acyclovir therapy who have positive CSF HSV PCR results within 48 hours prior to IV therapy completion, are not randomized.
Groups:
- Placebo: Identical to oral acyclovir suspension in appearance and taste. Volume is identical to the administration of active drug.
- Acyclovir: Oral suspension 300 mg/m^2/dose TID for 6 months.
Period: Overall Study
Arm/Group | Placebo | Acyclovir
Started | 14 | 15
Completed | 4 | 8
Not Completed | 10 | 7
Not completed — Lost to Follow-up | 0 | 1
Not completed — Non-compliant | 1 | 1
Not completed — Re-activation of Disease | 2 | 1
Not completed — Disruption of blinded study drug supply | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Acyclovir | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Customized [Median (Full Range); unit: days] | 15 (3.76) [5 to 55] | 15 (2.51) [2 to 35] | 15 (2.23) [2 to 55]
Age, Customized [Number; unit: participants]
  < = 28 days | 14 | 15 | 29
  Between 29 days and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 8 | 10 | 18
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28
  Canada | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Participants With Neurologic Impairment at 12 Months as Measured by a Bayley's Neuro-developmental Assessment.(Motor Scores)
Description: Motor scores of all participants completing 6 months of blinded therapy as measured by the Bayleys neuro-developmental assessment at 12 months. Scores are classified as the following: greater than or equal to 115 suggests accelerated performance; 85 - 114 suggests development within normal limits; 70 - 84 suggests mildly delayed development and less than or equal to 69 suggests significant delayed development.
Time Frame: At 12 months of life.
Population: Three of 4 subjects receiving placebo and completing 6 months of placebo, and 2 of 8 subjects receiving acyclovir and completing 6 months of acyclovir did not complete the 12 month Bayley's Neuro-developmental Assessment (motor score); therefore, 1 placebo subject and 6 acyclovir subjects are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo | Acyclovir
Number analyzed (Participants) | 1 | 6
Participants
  Number of participants with score of > or = 115 | 0 | 3
  Number of participants with score of 85 - 114 | 0 | 0
  Number of participants with score of 70 - 84 | 1 | 2
  Number of participants with score of < or = 69 | 0 | 1

2. Secondary Outcome: Detection of Herpes Simplex Virus (HSV) DNA in the Cerebrospinal Fluid (CSF) by Polymerase Chain Reaction (PCR) at Anytime During the Initial 12 Months of Life.
Description: Number of participants with positive herpes simplex virus (HSV) DNA by polymerase cahin reaction (PCR) in the cerebrospinal fluid of subjects assessed during the initial 12 months of life.
Time Frame: post randomization at 12 months
Measure: Number; unit: Participants
Arm/Group | Placebo | Acyclovir
Number analyzed (Participants) | 4 | 8
Participants
  Participants with at least 1 positive PCR | 0 | 0
  Participants with negative PCR or not done | 4 | 8

3. Secondary Outcome: Two or Fewer Episodes of Cutaneous Recurrence of HSV Disease Post-randomization During the Initial 12 Months of Life.
Description: Number of participants experiencing 2 or fewer HSV recurrences during the first 12 months of life as measured by assessments and reports at study visits.
Time Frame: post randomization - 12 months
Measure: Number; unit: participants
Arm/Group | Placebo | Acyclovir
Number analyzed (Participants) | 4 | 8
participants
  with < or = 2 recurrences of HSV | 4 | 7
  with > 2 recurrences of HSV | 0 | 1

4. Primary Outcome: Participants With Neurologic Impairment at 12 Months as Measured by a Bayley's Neuro-developmental Assessment.(Mental Scores)
Description: Mental scores of all participants completing 6 months of blinded therapy as measured by the Bayleys neuro-developmental assessment at 12 months. Scores are classified as the following: less than or equal to 115 suggests accelerated performance; 85 - 114 suggests development within normal limits; 70 - 84 suggests mildly delayed development and less than or equal to 69 suggests significant delayed development.
Time Frame: At 12 months of life.
Population: Two of 4 subjects receiving placebo and completing 6 months of placebo, and 2 of 8 subjects receiving acyclovir and completing 6 months of acyclovir did not complete the 12 month Bayley's Neuro-developmental Assessment(mental); therefore, 2 placebo subject and 6 acyclovir subjects are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo | Acyclovir
Number analyzed (Participants) | 2 | 6
Participants
  Number of participants score with > or = to 115 | 0 | 1
  Number of participants with score 85-114 | 1 | 1
  Number of participants with score 70-84 | 1 | 4
  Number of participants with < or = to 69 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | Acyclovir
Serious Adverse Events (participants affected / at risk) | 5/14 | 8/15
Other Adverse Events (participants affected / at risk) | 8/14 | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=14) | Acyclovir (N=15)
Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 3 (5)
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal refux (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Langerhans cell histocytosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Adenoiditis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex virus (Infections and infestations) | 1 (1) | 2 (2)
Lesion unspecified (Infections and infestations) | 2 (5) | 1 (1)
Neutropenia (Infections and infestations) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
RSV (Infections and infestations) | 0 (0) | 1 (1)
Near drowning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=14) | Acyclovir (N=15)
Decreased neutrophils (Blood and lymphatic system disorders) | 3 (6) | 5 (6)
Herpes simplex virus (Infections and infestations) | 2 (7) | 3 (3)
Infection ear (Infections and infestations) | 3 (4) | 6 (14)
Lesion-unspecified (Infections and infestations) | 5 (12) | 5 (7)
Upper respiratory infection (Infections and infestations) | 4 (4) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No